CLINICAL TRIAL: NCT06834620
Title: Impact of a Novel Primary School-based Physical Education Program on Physical and Motor Fitness of Malaysian Children: a Randomized Controlled Trial
Brief Title: School-Based Physical Education Program and Its Effects on Motor Fitness in Malaysian Children
Acronym: SPEP-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Naval Academy (Other)
Collaborators: Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia (Unknown)
Responsible Party: Principal Investigator, Gerasimos Grivas, Lecturer in Exercise Physiology, Hellenic Naval Academy, Hellenic Naval Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hellenic Naval Academy; PNURSP2025R424 (Other Grant/Funding Number: Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia)
Record Dates: First submitted 2025-02-09; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-01

CONDITIONS: Physical Fitness; Child Development; Exercise Intervention; Childhood Obesity; Physical Inactivity in Children
Keywords: Physical Education; Motor Fitness; Exercise Program
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rhythmic and Gymnastics-Based Exercise Group (Experimental): Participants in this arm received 80 sessions of a Rhythmic and Gymnastics-Based Physical Education Program (RGPEP) over an academic year. The program focused on rhythmic skills, gymnastics patterns, and movement-based activities designed to enhance motor and physical fitness.
  Interventions: Behavioral: Rhythmic and Gymnastic Activities-Based School Physical Education Program
- Control group (Active Comparator): Participants in this arm followed the standard Malaysian school physical education curriculum, which included 60 minutes of physical education and 30 minutes of health education per week, as prescribed by the Malaysian Ministry of Education.
  Interventions: Behavioral: Rhythmic and Gymnastic Activities-Based School Physical Education Program

INTERVENTIONS:
Behavioral: Rhythmic and Gymnastic Activities-Based School Physical Education Program — A structured, year-long school-based physical education program integrating rhythmic movements, gymnastics, and small equipment exercises designed to enhance motor and physical fitness. The program included 80 sessions (two per week) focusing on rhythmic activities such as twisting, partner balance, animal walks, tumbling, and rope exercises. The intervention aimed to improve strength, flexibility, agility, and cardiovascular endurance compared to traditional physical education classes.

SUMMARY:
The objective of this randomized controlled trial was to compare the effects of a standard school physical education program (SPEP) and a rhythmic and gymnastic activities-based school physical education program (RGPEP) on the physical and motor fitness parameters of Malaysian primary school children.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the impact of two distinct physical education programs on the physical and motor fitness of Malaysian primary school children. The intervention group participates in a rhythmic and gymnastic activities-based physical education program (RGPEP), designed to enhance balance, coordination, flexibility, and agility through structured, progressive activities. The control group follows the standard school physical education program (SPEP) in line with the national curriculum, which emphasizes general fitness and physical activity without specific rhythmic or gymnastic components.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 years at the time of enrollment.
* Both boys and girls.
* Regular school attendance during the academic year.
* No diagnosed health conditions or chronic diseases that could interfere with physical activity.
* Not involved in extracurricular sports activities outside the school environment.
* Not engaged in extra traveling to and from school on foot or by bicycle.
* Parents or legal guardians provided written informed consent.
* The child provided verbal assent to participate in the study.

Exclusion Criteria:

* Children missing more than 20% of scheduled physical education classes.
* Overweight children with a BMI ≥ 23 kg/m².
* Underweight children with a BMI < 18.5 kg/m².
* Children involved in regular sports training or participation in extracurricular sports activities during the intervention period.
* Children with any pre-existing medical conditions or injuries that could limit participation in physical activities.
* Children with developmental or motor impairments affecting their ability to perform the required fitness activities.
* Children on any medication that could interfere with their performance or physical fitness evaluation.

Ages: 8 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-02-14 (Actual); Primary Completion 2016-02-14 (Actual); Study Completion 2016-02-14 (Actual)

PRIMARY OUTCOMES:
Standing Broad Jump | Baseline (Month 0) and Post-Intervention (Month 12).
  The standing broad jump test measures lower body power in centimeters. Participants will perform a jump from a standing position, and the longest distance recorded will be used for analysis.
20-Meter Sprint | Baseline (Month 0) and Post-Intervention (Month 12).
  Sprint speed will be assessed using a 20-meter sprint test. The time taken (in seconds) to complete the distance will be recorded.
4 × 10-Meter Shuttle Run | Baseline (Month 0) and Post-Intervention (Month 12).
  Agility and speed will be measured using a 4 × 10-meter shuttle run test. Time to complete the test (in seconds) will be recorded.
Push-Ups | Baseline (Month 0) and Post-Intervention (Month 12).
  Upper body endurance will be assessed using the push-up test. The number of correctly executed push-ups performed will be recorded.
Sit and Reach Test | Baseline (Month 0) and Post-Intervention (Month 12).
  Flexibility will be assessed using the sit and reach test. The maximum reach distance (in centimeters) will be recorded.
Multistage Shuttle Run Test | Baseline (Month 0) and Post-Intervention (Month 12).
  Cardiovascular endurance will be measured using the multistage shuttle run test. VO₂max (mL/kg/min) will be estimated based on performance.

SECONDARY OUTCOMES:
Height | Baseline (Month 0) and Post-Intervention (Month 12).
  Standing height will be measured using a stadiometer and recorded in centimeters.
Weight | Baseline (Month 0) and Post-Intervention (Month 12).
  Body weight will be measured using a digital scale and recorded in kilograms.
Body Mass Index | Baseline (Month 0) and Post-Intervention (Month 12).
  BMI will be calculated as weight (kg) divided by height squared (m²).